CLINICAL TRIAL: NCT00610675
Title: Fifty-Two Weeks, Open Label Extension Trial to Evaluate Safety and Efficacy of Org 50081 in Outpatients With Chronic Primary Insomnia Who Completed Clinical Trial Protocol 176001 or 176002.
Brief Title: Fifty Two Week Extension Trial of Org 50081 (Esmirtazapine) in the Treatment of Insomnia (P05708)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05708; 176004
Record Dates: First submitted 2008-01-09; First posted 2008-02-08 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Insomnia
Keywords: Fifty two weeks; Open label; extension
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esmirtazapine (Experimental): One tablet of Esmirtazapine, 4.5 mg orally, daily for up to 52 weeks
  Interventions: Drug: Org 50081

INTERVENTIONS:
Drug: Org 50081 — One tablet daily

SUMMARY:
This trial is a 52-week, open-label extension trial to investigate safety and to explore efficacy of Org 50081 (Esmirtazapine) in participants who completed Protocol 176001 (P05706) (NCT00482612) or 176002 (P05707) (NCT00506389). Participants who have completed Protocol P05706 or P05707, and are willing to continue treatment with Esmirtazapine, can participate in Protocol 176004 (P05708) after signing informed consent.

ELIGIBILITY:
Inclusion Criteria:

* sign written informed consent after the scope and nature of the investigation have been explained to them, before any trial-related evaluations;
* completed Protocol P05706 or P05707;
* Have safety and efficacy assessments conducted per protocol P05706 or P05707.

Exclusion Criteria:

* clinically relevant electrocardiogram (ECG) abnormalities as judged by the investigator;
* clinically relevant abnormal laboratory values as judged by the investigator;
* any adverse event deemed relevant for exclusion in Protocol P05708 as judged by the investigator or,
* were significantly non compliant with protocol criteria and procedures of Protocol P05706 or P05707, as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2006-12-07 (Actual); Primary Completion 2009-08-17 (Actual); Study Completion 2009-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed base studies P05706 (NCT00482612) and P05707 (NCT00506389) were eligible to enroll in follow-up study P05708
Groups:
- Esmirtazapine: One tablet of Esmirtazapine, 4.5 mg daily for up to 52 weeks
Period: Overall Study
Arm/Group | Esmirtazapine
Started | 346
Treated | 342
Completed | 126
Not Completed | 220
Not completed — Untreated | 4
Not completed — Adverse Event | 67
Not completed — Insufficient Effect | 31
Not completed — Withdrawal by Subject | 28
Not completed — Reasons unrelated to trial | 27
Not completed — Lack of Compliance | 7
Not completed — Lost to Follow-up | 31
Not completed — Other reason (not specified) | 25

BASELINE CHARACTERISTICS:
Population: Participants treated with Esmirtazapine in Follow up trial P05708
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 342
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217
  Male | 125

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Description: An Adverse Event (AE) is any untoward occurrence in a participant who is administered any pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding) symptom, or disease temporarily associated with the use of an investigational medicinal product (IMP), whether or not it is related to the IMP.
Time Frame: Up to 57 weeks
Population: All subjects treated (AST) population consisting of all enrolled participants who received at least one dose of trial medication
Measure: Number; unit: Participants
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 342
Participants | 235

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: An Adverse Event (AE) is any untoward occurrence in a participant who is administered any pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding) symptom, or disease temporarily associated with the use of an IMP, whether or not it is related to the IMP.
Time Frame: Up to 52 weeks
Population: AST population consisting of all enrolled participants who received at least one dose of trial medication
Measure: Number; unit: Participants
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 342
Participants | 67

3. Secondary Outcome: Change From Baseline in Total Sleep Time at Week 52
Description: Total Sleep Time (TST) is a subjective time recorded by the participant in an electronic sleep diary in response to the question "How much time did you actually spend sleeping?". Baseline values were calculated by averaging baseline values from base trials P05706 and P05707. Data at baseline and at week 52 were collected every morning and evening for 7 consecutive days, and these data were then averaged. Missing values were imputed by the last observation carried forward (LOCF) method, where the last available assessments prior to the scheduled observation were averaged.
Time Frame: Baseline and Week 52
Population: AST participants who received at least one dose of trial medication and provided adequate data entries in their electronic sleep diary
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 290
Minutes
  Baseline (n= 290) | 331.7 (77.9)
  Change from Baseline (n= 285) | 73.0 (85.9)

4. Secondary Outcome: Change From Baseline in Sleep Latency at Week 52
Description: Sleep Latency (SL) is the time from when the participant went to bed up to the the time the participant actually fell asleep, recorded by the participant in an electronic sleep diary. Baseline values were calculated by averaging baseline values from base trials P05706 and P05707. Data at baseline and at week 52 were collected every morning and evening for 7 consecutive days, and these data were then averaged. Missing values were imputed by the LOCF method, where the last available assessments prior to the scheduled observation were averaged.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 290
Minutes
  Baseline (n= 290) | 70.9 (51.3)
  Change from Baseline (n= 285) | -24.5 (62.2)

5. Secondary Outcome: Change From Baseline in Wake Time After Sleep Onset at Week 52
Description: Wake time after sleep onset (WASO) is, if the planned waking time is on or after the time of final awakening, as follows: total time from falling asleep to the time of planned wake up minus the total sleep time. If the planned waking time is before the time of final awakening then WASO is as follows: total time from falling asleep to the time of actual final awakening minus the total sleep time. All times were recorded by the participant in an electronic sleep diary. Baseline values were calculated by averaging baseline values from base trials P05706 and P05707. Data at baseline and at week 52 were collected every morning and evening for 7 consecutive days, and these data were then averaged. Missing values were imputed by the LOCF method, where the last available assessments prior to the scheduled observation were averaged.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 290
Minutes
  Baseline (n= 290) | 85.0 (58.0)
  Change from Baseline (n= 285) | -34.8 (72.4)

6. Secondary Outcome: Change From Baseline in Number of Awakenings at Week 52
Description: Number of awakenings is a subjective number recorded by the participant in an electronic sleep diary. Baseline values were calculated by averaging baseline values from base trials P05706 and P05707. Data at baseline and at week 52 were collected every morning and evening for 7 consecutive days, and these data were then averaged. Missing values were imputed by the LOCF method, where the last available assessments prior to the scheduled observation were averaged.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 290
Awakenings
  Baseline (n= 290) | 2.0 (1.5)
  Change from Baseline (n= 285) | -0.7 (1.5)

7. Secondary Outcome: Change From Baseline in Quality of Sleep Scale at Week 52
Description: Quality of Sleep is a subjective number on a Visual Analog Scale recorded by the participant in an electronic sleep diary. The scale ranges from 0 to 100, where very poor is rated at 0, up to excellent, rated at 100. Baseline values were calculated by averaging baseline values from base trials P05706 and P05707. Data at baseline and at week 52 were collected every morning and evening for 7 consecutive days, and these data were then averaged. Missing values were imputed by the LOCF method, where the last available assessments prior to the scheduled observation were averaged.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 290
Units on a scale
  Baseline (n= 290) | 43.9 (17.9)
  Change from Baseline (n= 285) | 17.3 (22.0)

8. Secondary Outcome: Change From Baseline in Satisfaction With Sleep Duration Scale at Week 52
Description: Satisfaction with Sleep Duration is a subjective number on a Visual Analog Scale recorded by the participant in an electronic sleep diary. The scale ranges from 0 to 100, where very unsatisfied is rated at 0, up to fully satisfied, rated at 100. Baseline values were calculated by averaging baseline values from base trials P05706 and P05707. Data at baseline and at week 52 were collected every morning and evening for 7 consecutive days, and these data were then averaged. Missing values were imputed by the LOCF method, where the last available assessments prior to the scheduled observation were averaged.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 290
Units on a scale
  Baseline (n= 290) | 41.3 (17.8)
  Change from Baseline (n= 285) | 19.2 (22.2)

ADVERSE EVENTS:
Arm/Group | Esmirtazapine
Serious Adverse Events (participants affected / at risk) | 8/342
Other Adverse Events (participants affected / at risk) | 118/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine (N=342)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2)
Traumatic shock (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Victim of crime (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine (N=342)
Nasopharyngitis (Infections and infestations) | 26 (27)
Upper respiratory tract infection (Infections and infestations) | 20 (24)
Weight increased (Investigations) | 45 (50)
Somnolence (Nervous system disorders) | 44 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less